CLINICAL TRIAL: NCT07233499
Title: Evaluation of the Cardioprotective Effect of Nebivolol on Trastuzumab-Induced Cardiotoxicity in Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, May Ahmed Shawki, Associate professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHCLMSC200; NCI-323 (Other: National Cancer Institute- Cairo University- Egypt)
Record Dates: First submitted 2025-11-06; First posted 2025-11-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: Breast cancer; Nebivolol; trastuzumab; HER-2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Nebivolol

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebivolol (Experimental): Nebivolol group (28 patients): will receive nebivolol at a dose of 5 mg once daily (orally) during the whole period of receiving trastuzumab
  Interventions: Drug: Nebivolol 5 mg
- Control group (No Intervention): Control group (28 patients): will receive no intervention during the trastuzumab therapy

INTERVENTIONS:
Drug: Nebivolol 5 mg — nebivolol tablet 5 mg once daily
  Arms: Nebivolol

SUMMARY:
Breast cancer can be managed using chemotherapy, endocrine therapy and biological therapy. Treatment is determined and specified according to the characteristics of the tumor including overexpression of the human epidermal growth factor receptor (HER2). Previously patients who were diagnosed with HER2 positive breast cancer were considered of poor survival but after the discovery of trastuzumab, disease free survival among these patients was improved significantly.

Though trastuzumab has made great improvement in the treatment of breast cancer, it was identified to possess a major side effect which is cardiotoxicity . Cardiotoxicity that occurs with anticancer agents is usually manifested as left ventricular dysfunction (LVD) and overt heart failure (HF). LVD was defined as a decrease in cardiac LV ejection fraction (LVEF), that is either global or more severe in the septum, symptoms of congestive heart failure (CHF), associated signs of CHF including but not limited to S3 gallop, tachycardia or both and decline in LVEF of at least 5% to below 55% with accompanying signs or symptoms of CHF, or a decline in LVEF of at least 10% to below 55% without accompanying signs or symptoms.

Beta blockers have shown a cardioprotective effect against chemotherapy induced- cardiotoxicity.

Nebivolol is a third-generation beta blocker. It is highly selective to B1- adrenergic receptors. It also has peripheral vasodilating effect due to its effect on L-arginine/ nitric oxide pathway in the endothelium of blood vessels.

The dose of nebivolol given in the study was 5mg/day for the entire period of the study. Echo was done for all patients to determine the changes of left ventricular ejection fraction in patients in the treatment group and control group. The study concluded that nebivolol prevented the occurrence of anthracycline induced cardiotoxicity.

the current study will be the first clinical trial to evaluate the cardioprotective effect of nebivolol on trastuzumab-induced cardiotoxicity in breast cancer patients.

Aim of the work

Evaluation of the effect of Nebivolol on trastuzumab - induced cardiotoxicity in non-metastatic breast cancer patients by assessment of:

* Left ventricular ejection fraction.
* Cardiac biomarkers (troponin- Pro- BNP).
* Treatment safety.
* Patient quality of life (Using fact-B questionnaire)

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignancies that affect females around the world. According to the WHO, the number of females who were diagnosed with breast cancer in 2020 in Egypt was 22038 females. This number represents 32.4% of all women malignancies and 16.4% of all malignancies in Egypt (men and women).

Breast cancer can be managed using chemotherapy, endocrine therapy and biological therapy. Treatment is determined and specified according to the characteristics of the tumor including overexpression of the human epidermal growth factor receptor (HER2). Previously patients who were diagnosed with HER2 positive breast cancer were considered of poor survival but after the discovery of trastuzumab, disease free survival among these patients was improved significantly.

Trastuzumab is a humanized monoclonal antibody that was approved to treat HER2 positive breast cancer. Studies have shown that trastuzumab has improved the survival, reduced the mortality, reduced the recurrence and metastases rates in patients with HER2 positive breast cancer. Trastuzumab perform its tumor suppressive actions through different mechanisms that include activation of antibody-dependent cell-mediated cytotoxicity, inhibition of HER2 extracellular domain cleavage, disruption of HER2 receptor homodimerization and heterodimerization, abrogation of oncogenic cellular signaling and downregulation of angiogenesis and DNA repair pathways.

Though trastuzumab has made great improvement in the treatment of breast cancer, it was identified to possess a major side effect which is cardiotoxicity. Cardiotoxicity that occurs with anticancer agents is usually manifested as left ventricular dysfunction (LVD) and overt heart failure (HF). LVD was defined as a decrease in cardiac LV ejection fraction (LVEF), that is either global or more severe in the septum, symptoms of congestive heart failure (CHF), associated signs of CHF including but not limited to S3 gallop, tachycardia or both and decline in LVEF of at least 5% to below 55% with accompanying signs or symptoms of CHF, or a decline in LVEF of at least 10% to below 55% without accompanying signs or symptoms.

According to a study conducted by Mohan et al in 2016, It was shown that treatment with trastuzumab leads to inhibition of HER2 signaling and phosphorylation of HER1-Y845/HER2-Y1248 and the activation of Erk. All this consequently leads to upregulation of the mTOR-Ulk1 pathway to mediate inhibition of autophagy in cardiomyocytes. This was clearly shown by the decrease in expression levels of LC3 I/II and increase in p62 after trastuzumab treatment. Studies has shown that inhibition of autophagy by autophagy inhibitor (3-methyladenine) leads to accumulation of damaged mitochondria and increase the concentration of mitochondrial ROS and thus accumulation of toxic reactive oxygen species (ROS) in human cardiomyocytes which can lead to oxidative damage and cardiotoxicity.

Beta blockers have been used to treat ischemic heart disease due to their negative chronotropic and inotropic properties thus inducing a decrease in myocardial consumption of oxygen and nutrients allowing better balance between nutritional needs and blood flow. Recent studies have proved that not all beta blockers have equal effect as their intercellular mechanisms of action are different. Beta blockers have shown a cardioprotective effect against chemotherapy induced- cardiotoxicity.

Nebivolol is a third-generation beta blocker. It is highly selective to B1- adrenergic receptors. It also has peripheral vasodilating effect due to its effect on L-arginine/ nitric oxide pathway in the endothelium of blood vessels. Nitric oxide is a paracrine factor derived from the endothelial cells and alleviate ROS mediated oxidative damage. Nebivolol activates the endothelial nitric oxide system and increases nitric oxide release through activation of the beta 3 adrenergic receptors in endothelium cells. The release of nitric oxide causes peripheral vasodilation, an increase in the myocardial compliance and an inhibition of inotropic effect of sympathetic stimulation. Nebivolol also decreases the nitric oxide break down and increases its bioavailability. All these effects of nebivolol on nitric oxide lead to a decrease in cardiac load, an enhanced cardiac filling and a protection of myocardium.

In a meta-analysis of 12 clinical trials, it was found that there was a great decrease in reactive oxygen species (ROS) concentration in endothelial cells exposed to oxidative stress in patients who were taking nebivolol in comparison to other patients who were receiving other beta blockers. Besides, it was found that the decrease of basal and stimulated nitric oxide because of oxidative stress is less in patients taking nebivolol compared to other patients. This all shows that nebivolol has antioxidant properties which reduce oxidative stress and affects organs damage.

The animal study which is conducted in 2018 to assess the Protective effect of nebivolol on doxorubicin-induced cardiotoxicity in rats. The specimens were examined using H + E and Masson's trichrome, caspase 3, endothelial nitric oxide synthase (eNOS), inducible nitric oxide synthase (iNOS) and tumor necrosis factor factor-α (TNF-α). The mean area percentage of collagen fiber content, caspase-3, eNOS, iNOS and TNF-α immunoactivities was measured. Doxorubicin-treated group showed marked myocyte distortion and fragmentation, congestion and cytoplasmic lysis in most fibers. These changes were less intense in the nebivolol-treated group. The study concluded that nebivolol exerted a significant protective effect from doxorubicin toxicity. The protective effect appears to be mediated mainly through caspase-3, eNOS, iNOS and TNF-α modulation.

Cochera and his colleagues conducted a study in 2018 to assess the effect of nebivolol treatment in the prevention of anthracyclines induced cardiotoxicity. The dose of nebivolol given in the study was 5mg/day for the entire period of the study. Echo was done for all patients to determine the changes of left ventricular ejection fraction in patients in the treatment group and control group. The study concluded that nebivolol prevented the occurrence of anthracycline induced cardiotoxicity.

the current study will be the first clinical trial to evaluate the cardioprotective effect of nebivolol on trastuzumab-induced cardiotoxicity in breast cancer patients.

Aim of the work

Evaluation of the effect of Nebivolol on trastuzumab - induced cardiotoxicity in non-metastatic breast cancer patients by assessment of:

* Left ventricular ejection fraction.
* Cardiac biomarkers (troponin- Pro- BNP).
* Treatment safety.
* Patient quality of life (Using fact-B questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Newly diagnosed with early or locally advanced HER2 positive breast cancer.
* Normal baseline LVEF (˃50%)
* Planned to receive HER2-directed therapies as newadjuvant or adjuvant.

Exclusion Criteria:

* Elderly patients( ˃65 years).

  * Primary tumors other than breast cancer.
  * Pregnancy and breast feeding.
  * Currently using cardioprotective drugs e.g.: ACEI, CCB, ARBs and another beta blocker.
  * Presence of diagnosed cardiomyopathy currently or in initial evaluation.
  * Patients with ischemic heart disease.
  * Contraindication for treatment with beta blockers.
  * Patients with hypersensitivity to nebivolol.
  * Poorly echogenic patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 56 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Left ventricular ejection fraction by Echocardiography | 12 months
  Echo will be done at baseline (before start of trastuzumab) and every 3 months during receiving trastuzumab to evaluate the reduction in the left ventricular ejection fraction and overall cardiac function

SECONDARY OUTCOMES:
II-Evaluation of cardiac biomarkers. | 12 months
  Serum and plasma samples will be withdrawn from every patient at baseline, before surgery , after surgery and at the end of the study. Serum samples for evaluation of troponin and plasma samples for evaluation of pro-BNP. The samples will be stored at -20 till analysis.
Number of participants with treatment-related adverse events | 12 months.
  Patients 'blood samples will be taken at baseline, 6 months and 12 months to check their liver functions, kidney functions and CBC. Nebivolol side effects will be followed up during regular phone calls with the patients every two weeks. the number of participants with adverse events will be recorded
Evaluation of Quality of Life. | 12 months
  ● The quality of life will be assed using Functional assessment of cancer therapy-Breast (FACT-B) at baseline, after 6 months and at the end of the study. the questionnaire assesses functional, social , physical and emotional well being. The score ranges from 0-148 with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute- Cairo University- Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No